CLINICAL TRIAL: NCT07315984
Title: Multi-Modal Digital Monitoring of Disease Symptoms Huntington's Disease
Acronym: BioDigit HD-02
Status: Not yet recruiting | Type: Observational
Sponsor: BioSensics (Industry)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); University of Rochester - CHeT/CTCC (Unknown); Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: BioDigit HD-02; 1R44TR005381-01A1 (NIH)
Record Dates: First submitted 2025-12-30; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Huntington Disease
Keywords: huntington disease; wearable sensors; digital health
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hungtinton's Disease: Participants with clinical diagnosis of HD
- Age-matched healthy adults: Age-matched healthy adults. Clinically assessed to be in good health, with no evidence of neurological disorders that could cause involuntary movements or gait disturbances.

SUMMARY:
The objective of the study is to validate the use of wearable sensors and digital health technologies for monitoring disease activity in Huntington's Disease (HD). Healthy subjects, as well as subjects with documented diagnosis of HD will be screened and recruited at University of Rochester Medical Center and Vanderbilt University Medical Center to participate in this 12-month observational study. There will be a total of 5 visits every approximately 3 months.

In each study visit, participants will complete several Patient Reported Outcomes (PROs), Clinical Reported Outcomes, complete a series of Digital Assessments (Speech, Cognitive, Motor, and Finger Tapping). Participants will be provided with a pendant, wrist, and ankle sensors to monitor their daily physical activities for 7 days after each study visit. Participants will also be provided with a tablet to complete digital assessments (Speech, Cognitive, Motor, and Finger Tapping) on monthly basis at home.

DETAILED DESCRIPTION:
HD is a devastating inherited neurological disorder that causes progressive nerve degeneration in the brain. HD is characterized by multifaceted symptomatology including motor, cognitive, and psychiatric symptoms, which begin insidiously and progress over many years. The principal means of measuring gross motor and speech impairment in HD is the Unified Huntington's Disease Rating Scale (UHDRS). Although valuable, the scale is subjective and categorical and requires significant training to administer correctly. Quantitative motor (Q-motor) tests have helped reduce subjectivity and improve sensitivity of motor assessments in HD. Q-Motor assessments have demonstrated utility in tracking longitudinal progression of motor impairment and as a supplemental measure in clinical trials. Likewise, force-sensitive insoles, video motion analysis systems, and pressure-sensitive walking mats have been utilized to objectively measure impaired gait in HD. However, these gait-measuring technologies and Q-Motor assessments must be administered in clinic by trained personnel. Similarly, the Montreal Cognitive assessment (MoCA) and Mini-mental State Examination, are often used to measure cognitive decline. However, these tests need to be administered by trained professionals and have limited ability to detect subtle changes in cognitive performance over time. Furthermore, measures are conducted infrequently, typically in a clinic setting, and may not be an accurate representation of an individual's true cognitive status.

There is currently no cure which can halt, slow or reverse the progression of the disease. The key challenge in development of new therapeutics in HD and other neurological disorders is that the current way of assessing the disease is largely subjective and requires in-person, in-clinic assessments. Digital measures, like the proposed solution can provide objective, real-world assessments of how individuals are functioning.

Wearable sensors and digital health technologies that can detect motor, speech, and cognitive abnormalities can provide insight into the phase of clinical disease onset. Given that gene positive premanifest stage of HD can take up to several years before the onset of symptomatic disease, the subtle changes in these biomarkers in the early stage of HD provide an opportune window to apply disease-modifying treatment that could potentially slow down or prevent the progression of the disease

Thus, a system that can objectively, sensitively, and frequently monitor multiple clinical domains (motor, speech and cognitive function) is necessary to understand the pattern of evolving motor, speech and cognitive abnormalities in individuals with prodromal HD, and for identification of endpoint measures for therapeutic trials.

This observational study will follow participants over 12 months. Healthy subjects, as well as subjects with documented diagnosis of HD will be screened and recruited at University of Rochester Medical Center and Vanderbilt University Medical Center. In addition to standard clinical assessments, the study will leverage BioDigit HD to collect wearable and digital health data from participants in at the study site and their home environments.

A key objective of the project is to measure changes in disease symptoms using patient reported outcomes (PROs), clinical reported outcomes, and digital measures in individuals with HD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 25-65 years
* For HD participants: Genetically diagnosed with HD
* Fluent in English (able to speak and read).
* Ambulatory without the need for a walking aid.
* Able to independently perform all study activities safely, as determined by the investigator.
* Willing and able to provide informed consent and comply with all study procedures.

For control participants:

* Male or female, aged 25-65 years
* Clinically assessed to be in good health, with no evidence of neurological disorders that could cause involuntary movements or gait disturbances

Exclusion Criteria:

* Diagnosis of juvenile-onset HD.
* Individuals who are non-ambulatory.
* Individuals with a neurological, medical, or psychiatric condition that, in the investigator's judgment, would interfere with safe participation in study activities.
* Montreal Cognitive Assessment (MoCA) score of 18 or lower
* Pregnant individuals, due to potential changes in gait and physical activity during pregnancy.
* Cannot be enrolled into a blinded intervention trial at baseline.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with clinical diagnosis of HD, and healthy age-matched controls
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in daily walking duration during activities of daily living from baseline to 12 months as measured by the PAMSys pendant | 12 months
  Daily walking duration (hours) will be measured by the PAMSys pendant. PAMSys is a FDA-listed Class II wearable device for measuring physical activity and posture during activities of daily living.
  PAMSys will be worn for 1 week after the baseline, 3 month, 6 month, 9 month, and 12 month visits.
Change in daily number of sit to stand transitions (count) during activities of daily living from baseline to 12 months as measured by the PAMSys pendant. | 12 months
  Daily number of sit to stand transitions will be measured by the PAMSys pendant. PAMSys is a FDA-listed Class II wearable device for measuring physical activity and posture during activities of daily living.
  PAMSys will be worn for 1 week after the baseline, 3 month, 6 month, 9 month, and 12 month visits.

SECONDARY OUTCOMES:
Change in scores of Unified Huntington's Disease Rating Scale (UHDRS) from baseline to 12 months | 12 months
  A clinical tool used to assess motor, cognitive, and behavioral symptoms in individuals with Huntington's disease (HD).
  There are 5 parts to UHDRS
  1. Total Motor Score: Scores range from 0 to 124. Higher scores represent a worse outcome.
  2. Total Functional Capacity: Scores range from 0 to 13. Lower scores represent a worse outcome.
  3. Behavioral Assessment: Scores range from 0 to 88. Higher scores represent a worse outcome.
  4. Cognitive Assessments: Inclues Stroop test, Verbal Fluency, and Symbol Digit Modalities Test. Lower scores represent a worse outcome.
Change in intelligibility when reading a standard Rainbow passage from baseline to 12 months as measured by BioDigit Speech | 12 months
  Speech data will be collected from participants while reading a standard Rainbow passage on a monthly basis for 12 months. BioDigit Speech, and automatic speech analysis software, will be used to analyze the collected speech data to calculate intelligibility of speech during reading a standard Rainbow passage.
Change in walking speed during activities of daily living from baseline to 12 months as measured by the PAMSys Ankle sensor | 12 months
  median, 90 percentile and 96 percentile stride velocity (m/s) will be measured by the PAMSys Ankle sensor. PAMSys Ankle sensor will be worn for 1 week after the baseline, 3 month, 6 month, 9 month, and 12 month visits.
Change in cadence during activities of daily living from baseline to 12 months as measured by the PAMSys pendant | 12 months
  Median, 90 percentile and 96 percentile cadence (steps/min) will be measured by the PAMSys pendant. PAMSys pendant will be worn for 1 week after the baseline, 3 month, 6 month, 9 month, and 12 month visits.
Change in the Montreal Cognitive assessment (MoCA) score | 12 months
  The MoCA will be assessed from participants during baseline, 3 month, 6 month, 9 month and 12 month visits.

OTHER OUTCOMES:
Change in tapping rate (number of taps per minute) from baseline to 12 months as measured by the BioDigit Clinic and BioDigit Home tablets | 12 months
  Finger tapping test will be collected from participants on a monthly basis for 12 months.
Change in daily number of hand goal-directed movements during activities of daily living from baseline to 12 months as measured by the PAMSys ULM wrist sensor | 12 months
  PAMSys ULM wrist sensor measures goal directed movements of the hand during activities of daily living. PAMSys ULM wrist sensors will be worn for 1 week after the baseline, 3 month, 6 month, 9 month, and 12 month visits.
Change in the Verbal Fluency test score | 12 months
  Verbal fluency test data will be collected at baseline, 3 month, 6 month, 9 month and 12 month visits.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Rochester Medical Center, Rochester, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No